CLINICAL TRIAL: NCT02905357
Title: Heart Attack Research Program- Imaging Study
Acronym: HARP
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 16-01104-2
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Imaging
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood collection in platelet substudy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MINOCA: OCT and CMR imaging
  Interventions: Device: OCT
- MI-CAD: Screen failures with MI found to have obstructive CAD. Limited data collection for comparison to MINOCA cohort.
  Interventions: Other: CMR

INTERVENTIONS:
Device: OCT — Optical Coherence Tomography (OCT): Intracoronary imaging for amount and type of plaque as well as plaque rupture, ulceration, dissection and/or thrombosis.
  Groups: MINOCA
Other: CMR — Cardiac Magnetic Resonance Imaging (CMR): MRI of the heart to identify areas of infarction (damage) and/or edema (swelling).
  Groups: MI-CAD

SUMMARY:
The HARP study is a multi-center, diagnostic observational study employing standardized imaging protocols in patients with MINOCA (MI with Non Obstructive Coronary Arteries) to determine the underlying diagnosis in each participant. Participants will be followed for recurrent clinical events, every 6 months, for a maximum of 10 years.

DETAILED DESCRIPTION:
HARP is a multi-center, observational study which enrolls men and women with MI who are referred for cardiac catheterization. Eligible participants with MINOCA (defined as no stenosis of >50% in any major epicardial vessel) will undergo optical coherence tomography (OCT) at the time of diagnostic angiography and cardiac magnetic resonance imaging (CMR).

Participants will also have the option to enroll in the HARP-Platelet Sub-Study.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic symptoms compatible with diagnosis of MI, such as chest pain or anginal equivalent symptoms at rest or new onset exertional anginal equivalent symptoms
* Objective evidence of MI (either or both of the following):

  * Elevation of troponin to above the laboratory upper limit of normal
  * ST segment elevation of ≥1mm on 2 contiguous ECG leads
* Willing to provide informed consent and comply with all aspects of the protocol
* Age ≥ 21 years

Exclusion Criteria:

* Stenosis ≥50% of any major epicardial vessel on invasive angiography, as determined by the angiographer at the time of clinically ordered cardiac catheterization
* History of known obstructive coronary artery disease at angiography, including history of percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
* Recent use of vasospastic agents, such as cocaine, triptans, or ergot alkaloids (≤1 month)
* Alternate explanation for troponin elevation, such as hypertensive urgency, acute exacerbation of heart failure, chronic elevation due to kidney disease, pulmonary embolism, cardiac trauma
* Coronary dissection apparent on angiography
* Excessive coronary tortuosity which, in the angiographer's opinion, increases the risks of OCT
* eGFR<45 or contraindication to additional contrast needed for OCT in the opinion of the angiographer or treating physician
* Contraindication to MRI (including but not limited to ferromagnetic implants)
* Pregnancy
* Thrombolytic therapy for STEMI (qualifying event)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with MI and no coronary stenosis of 50% or greater on angiography, consecutive.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with MINOCA who have plaque disruption (any of the following: rupture, erosion, calcified nodule with thrombosis) | 1 week

SECONDARY OUTCOMES:
Proportion of patients with MINOCA who have spontaneous coronary dissection. | 1 week
Proportion of patients with MINOCA who have late gadolinium enhancement and/or myocardial edema | 1 week
Correlation of the presence and location of myocardial abnormalities on CMR with presence and location of plaque disruption on OCT among women with MINOCA. | 1 week
Proportion of patients for whom an etiology can be clearly identified after combining OCT and CMR. | 1 week
Area under curve of clinical prediction model for plaque disruption on OCT in patients with MINOCA. | 1 week

OTHER OUTCOMES:
Composite clinical endpoint: Death, unstable angina, stroke, recurrent MI, catheterizations and revascularization, other cardiac hospitalization. | 10 years
  components of composite will also be examined
Perceived stress | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Harmony R Reynolds, MD, Principal Investigator — NYU Langone Medical Center
Locations (19):
- United States (15):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC San Diego Medical Center, San Diego, California
  - Stanford University, Stanford, California
  - University of Florida Medical Center, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - NYU Winthrop, Mineola, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Seton Heart (Ascension) Univeristy of Austin, Texas, Austin, Texas
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - University of Calgary, Calgary

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared after the end of the study.

REFERENCES:
- [Derived] Arabadjian M, Duberstein ZT, Sperber SH, Kaur K, Kalinowski J, Xia Y, Hausvater A, O'Hare O, Smilowitz NR, Dickson VV, Zhong H, Berger JS, Hochman JS, Reynolds HR, Spruill TM. Role of Resilience in the Psychological Recovery of Women With Acute Myocardial Infarction. J Am Heart Assoc. 2023 Apr 18;12(8):e027092. doi: 10.1161/JAHA.122.027092. Epub 2023 Apr 7. PMID 37026542
- [Derived] Usui E, Matsumura M, Smilowitz NR, Mintz GS, Saw J, Kwong RY, Hada M, Mahmud E, Giesler C, Shah B, Bangalore S, Razzouk L, Hoshino M, Marzo K, Ali ZA, Bairey Merz CN, Sugiyama T, Har B, Kakuta T, Hochman JS, Reynolds HR, Maehara A. Coronary morphological features in women with non-ST-segment elevation MINOCA and MI-CAD as assessed by optical coherence tomography. Eur Heart J Open. 2022 Sep 30;2(5):oeac058. doi: 10.1093/ehjopen/oeac058. eCollection 2022 Sep. PMID 36225342
- [Derived] Reynolds HR, Kwong RY, Maehara A, Smilowitz NR. Response by Reynolds et al to Letters Regarding Article, "Coronary Optical Coherence Tomography and Cardiac Magnetic Resonance Imaging to Determine Underlying Causes of Myocardial Infarction With Nonobstructive Coronary Arteries in Women". Circulation. 2021 Sep 21;144(12):e209-e210. doi: 10.1161/CIRCULATIONAHA.121.055516. Epub 2021 Sep 20. No abstract available. PMID 34543066
- [Derived] Reynolds HR, Maehara A, Kwong RY, Sedlak T, Saw J, Smilowitz NR, Mahmud E, Wei J, Marzo K, Matsumura M, Seno A, Hausvater A, Giesler C, Jhalani N, Toma C, Har B, Thomas D, Mehta LS, Trost J, Mehta PK, Ahmed B, Bainey KR, Xia Y, Shah B, Attubato M, Bangalore S, Razzouk L, Ali ZA, Merz NB, Park K, Hada E, Zhong H, Hochman JS. Coronary Optical Coherence Tomography and Cardiac Magnetic Resonance Imaging to Determine Underlying Causes of Myocardial Infarction With Nonobstructive Coronary Arteries in Women. Circulation. 2021 Feb 16;143(7):624-640. doi: 10.1161/CIRCULATIONAHA.120.052008. Epub 2020 Nov 14. PMID 33191769